CLINICAL TRIAL: NCT01144208
Title: The Influence of Local Bone Status on Complications After Surgical Treatment of Distal Radius Fractures
Status: Completed | Type: Observational
Sponsor: AO Clinical Investigation and Publishing Documentation (Other)
Responsible Party: Dr D. Rikli, Universitätsspital Basel, Behandlungszentrum Bewegungsapparat BZB, Spitalstrasse 21, CH-4031 Basel, Switzerland
Organization: AO Innovation Translation Center (Other)
Other Study IDs: FFOB-Rad
Record Dates: First submitted 2010-06-14; First posted 2010-06-15 (Estimated); Last update posted 2010-06-16 (Estimated); Status verified 2010-06

CONDITIONS: Distal Radius Fractures; Poor Bone Quality; Treatment Complications
Keywords: Radius fracture; Adverse effects; Wrist; Postoperative complications; Colles' fracture; Intraoperative complications; Osteoporosis; Dual-energy x-ray absorptiometry (DXA); Bone Density
MeSH Terms: conditions — Wrist Fractures; Radius Fractures; Postoperative Complications; Colles' Fracture; Intraoperative Complications; Osteoporosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate if poor bone quality increases the risk of specific types of treatment complications in patients with distal radius fractures treated with open reduction and Locking Compression Plates(LCP).

DETAILED DESCRIPTION:
Despite fractures of the wrist being widely regarded as "fragility fractures", there is good evidence that they are caused by diminished Bone Mineral Density (BMD) and that a low BMD value predicts a higher fracture risk at the distal radius. Both measurements of areal BMD with DXA and volumetric BMD with peripheral Quantitative Computer Tomography (pQCT)showed a lower BMD in women with Colles' fractures. Thus, Colles' fractures can be recognized as a good indication of underlying osteoporosis. High resolution peripheral Quantitative Computer Tomography at the distal radius will be evaluated in a subset of patients.

Clinical experts are concerned that osteoporosis increases the risk for poor outcomes and complication rates in surgical patients with osteoporosis. However, this has not yet been confirmed in clinical studies. It is important to investigate this question in order to correctly advise clinicians and patients and possibly develop tailored approaches for treatment of osteoporotic patients with distal radius fractures.

ELIGIBILITY:
Inclusion Criteria:

* Radiologically confirmed closed fracture (within 7 days) of the distal radius
* Primary fracture treatment with a volar LCP 2.4 mm
* Age equal greater 50 and equal younger 90 years
* Willing and able to give written informed consent to participate in the study
* Willing and able to participate in the study follow-ups according to the CIP
* Willing and able to comply with the post-operative management program
* Able to understand and read country national language at an elementary level

Exclusion Criteria:

* Fracture of ulna (except an associated fracture of the ulnar styloid process)
* Open distal radius fracture
* Concomitant contralateral radius fracture
* Previous distal radius fracture on either side after the age of 25 years
* Time to operation > 7 days
* Polytrauma
* Regular systemic therapy with corticosteroids due to chronic disease
* Legal incompetence
* Patient received radio- or chemotherapy prior to, during, or within the last year
* Currently active cancer
* Recent history of substance abuse (i.e recreational drugs, alcohol)
* Prisoner
* Currently involved in a pharmaceutical study
* Has a disease process that would preclude accurate evaluation (e.g. neuromuscular or rheumatic disease, significant psychiatric or metabolic disorders)

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: participating clinics will identify all eligible patients who meet the inclusion and exclusion
Sampling Method: Probability Sample
Enrollment: 244 (Actual)
Dates: Start 2007-02; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Local bone quality-related complication | From enrollment to 12 months postoperative
  The qualifying events are those involving either directly the local bone and fracture or the implant and its surgical application whether they are anticipated or not.

SECONDARY OUTCOMES:
Bone mineral density at contralateral distal radius by DXA | until 6 weeks postoperative
  Local bone status will comprise BMD and BMC of the contralateral side. The absolute values for BMD and BMC will be provided as well as the deviations to the T-score according to the manufacturer's reference collective.
Occurence of any complication | Baseline
  To capture any complication that occured. A complication is defined as any occurrence or deviation from the normal treatment or outcome, regardless of whether it has any relationship with the treatment or product under investigation.
Occurence of any complication | 6 weeks
  To capture any complication that occured. A complication is defined as any occurrence or deviation from the normal treatment or outcome, regardless of whether it has any relationship with the treatment or product under investigation.
Occurence of any complication | 3 months
  To capture any complication that occured. A complication is defined as any occurrence or deviation from the normal treatment or outcome, regardless of whether it has any relationship with the treatment or product under investigation.
Occurence of any complication | 12 months
  To capture any complication that occured. A complication is defined as any occurrence or deviation from the normal treatment or outcome, regardless of whether it has any relationship with the treatment or product under investigation.
Range of motion | 6 weeks
  The bilateral range of motion will be measured by clinical examination as follows:
  * Dorsal extension / palmar flexion
  * Wrist ulnar abduction / radial abduction
  * Forearm supination / pronation
Range of motion | 3 months
  The bilateral range of motion will be measured by clinical examination as follows:
  * Dorsal extension / palmar flexion
  * Wrist ulnar abduction / radial abduction
  * Forearm supination / pronation
Range of motion | 12 months
  The bilateral range of motion will be measured by clinical examination as follows:
  * Dorsal extension / palmar flexion
  * Wrist ulnar abduction / radial abduction
  * Forearm supination / pronation
Grip strength | 6 weeks
  For the grip strength, the average value of three successive measurements with a Jamar dynamometer will be calculated as percentage of the contralateral, healthy side.
Grip strength | 3 months
  For the grip strength, the average value of three successive measurements with a Jamar dynamometer will be calculated as percentage of the contralateral, healthy side.
Grip strength | 12 months
  For the grip strength, the average value of three successive measurements with a Jamar dynamometer will be calculated as percentage of the contralateral, healthy side.
Patient self-assessment of wrist function questionnaire (PRWE) | Baseline
  PRWE was developed to rate wrist-related pain and disability in functional activities. This provides a score from 0-100, where higher scores indicate greater pain and disability.
Patient self-assessment of hand function with the PRWE | 6 weeks
  PRWE was developed to rate wrist-related pain and disability in functional activities. This provides a score from 0-100, where higher scores indicate greater pain and disability.
Patient self-assessment of hand function with the PRWE | 3 months
  PRWE was developed to rate wrist-related pain and disability in functional activities. This provides a score from 0-100, where higher scores indicate greater pain and disability.
Patient self-assessment of hand function with the PRWE | 6 months
  PRWE was developed to rate wrist-related pain and disability in functional activities. This provides a score from 0-100, where higher scores indicate greater pain and disability.
Patient self-assessment of hand function with the PRWE | 12 months
  PRWE was developed to rate wrist-related pain and disability in functional activities. This provides a score from 0-100, where higher scores indicate greater pain and disability.
Disabilities of the arm, shoulder and hand questionnaire (DASH) | Baseline
  The disability of the arm, shoulder and hand (DASH) questionnaire is an upper extremity specific outcome measure. The main part of the DASH is a 30-item disability/symptom scale concerning the patient's health status during the preceding week. The scores for all items are then used to calculate a scale score ranging from 0 (no disability) to 100 (most severe disability).
Disabilities of the arm, shoulder and hand questionnaire (DASH) | 6 weeks
  The disability of the arm, shoulder and hand (DASH) questionnaire is an upper extremity specific outcome measure. The main part of the DASH is a 30-item disability/symptom scale concerning the patient's health status during the preceding week. The scores for all items are then used to calculate a scale score ranging from 0 (no disability) to 100 (most severe disability).
Disabilities of the arm, shoulder and hand questionnaire (DASH) | 3 months
  The disability of the arm, shoulder and hand (DASH) questionnaire is an upper extremity specific outcome measure. The main part of the DASH is a 30-item disability/symptom scale concerning the patient's health status during the preceding week. The scores for all items are then used to calculate a scale score ranging from 0 (no disability) to 100 (most severe disability).
Disabilities of the arm, shoulder and hand questionnaire (DASH) | 12 months
  The disability of the arm, shoulder and hand (DASH) questionnaire is an upper extremity specific outcome measure. The main part of the DASH is a 30-item disability/symptom scale concerning the patient's health status during the preceding week. The scores for all items are then used to calculate a scale score ranging from 0 (no disability) to 100 (most severe disability).
Health-related quality of life (EQ-5D) | Baseline
  EQ-5D is a standardised instrument for use as a measure of health outcome.It has five items with a three-point categorical response scale (no problems, some/moderate problems, extreme problems. A unique EQ-5D health state is defined by combining 1 level from each of the 5 dimensions.
Health-related quality of life (EQ-5D) | 6 weeks
  EQ-5D is a standardised instrument for use as a measure of health outcome.It has five items with a three-point categorical response scale (no problems, some/moderate problems, extreme problems. A unique EQ-5D health state is defined by combining 1 level from each of the 5 dimensions.
Health-related quality of life (EQ-5D) | 3 months
  EQ-5D is a standardised instrument for use as a measure of health outcome.It has five items with a three-point categorical response scale (no problems, some/moderate problems, extreme problems. A unique EQ-5D health state is defined by combining 1 level from each of the 5 dimensions.
Health-related quality of life (EQ-5D) | 6 months
  EQ-5D is a standardised instrument for use as a measure of health outcome.It has five items with a three-point categorical response scale (no problems, some/moderate problems, extreme problems. A unique EQ-5D health state is defined by combining 1 level from each of the 5 dimensions.
Health-related quality of life (EQ-5D) | 12 months
  EQ-5D is a standardised instrument for use as a measure of health outcome.It has five items with a three-point categorical response scale (no problems, some/moderate problems, extreme problems. A unique EQ-5D health state is defined by combining 1 level from each of the 5 dimensions.
High resolution pQCT of contralateral distal radius | within 6 weeks after surgery
  High-resolution pQCT of the contralateral side with an XTremeCT will be performed in a subset of patients in Zürich. To obtain the bone mineral content the CT values will be calibrated with the help of a phantom in hydoxyapatite (HA) densities in mg HA/cm3. The relation of bone volume to tissue volume will be calculated as BV/TV. These values will be analyzed separately.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel A Rikli, PD, Principal Investigator — Universitätsspital Basel
Locations (11):
- Massachusetts General Hospital, Boston, Massachusetts, United States
- Universitätsklinik für Unfallchirurgie, Graz, Styria, Austria
- Germany (3):
  - Klinikum rechts der Isar der TU Muenchen, Munich, Bavaria
  - Ev. Diakoniewerk Friederikenstift, Hanover, Lower Saxony
  - Campus Virchow-Klinikum, Charité, Berlin, State of Berlin
- C.T.O. Azienda Ospedaliera Careggi, Florence, Tuscany, Italy
- Singapore General Hospital, Singapore, Singapore, Singapore
- Switzerland (4):
  - Universitätsspital Basel, Basel, Basel
  - Kantonsspital, Lucerne, Canton of Lucerne
  - Kantonsspital Winterthur, Winterthur, Canton of Zurich
  - Stadtspital Triemli, Zurich, Canton of Zurich

REFERENCES:
- [Derived] Goldhahn S, Kralinger F, Rikli D, Marent M, Goldhahn J. Does osteoporosis increase complication risk in surgical fracture treatment? A protocol combining new endpoints for two prospective multicentre open cohort studies. BMC Musculoskelet Disord. 2010 Nov 9;11:256. doi: 10.1186/1471-2474-11-256. PMID 21062463
- See also: Non profit organization dedicated to improving the care of patients with musculoskeletal injuries and their sequelae through research, development, education and quality assurance in the principles, practice, and result of fracture treatment. — http://www.aofoundation.org